CLINICAL TRIAL: NCT01796093
Title: Comparison of Digoxin and Ivabradine in Heart Failure With Preserved Systolic Function.
Brief Title: Digoxin Versus Ivabradine in Heart Failure With Preserved Systolic Function
Acronym: DIGvsIVA
Status: Completed | Type: Observational
Sponsor: Cocco, Giuseppe, M.D. (Individual)
Collaborators: Cardiology Office, Rheinfelden, Switzerland (Other)
Responsible Party: Principal Investigator, Cocco G., M.D., M.D., FESC, Cocco, Giuseppe, M.D.
Other Study IDs: GC&PJ-Dig-Iva-2009-2012; Cocco G, M.D. (Other Grant/Funding Number: Cocco G, MD)
Record Dates: First submitted 2012-09-05; First posted 2013-02-21 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Heart Failure; Atrial Fibrillation
Keywords: Digoxin; Ivabradine; Cardiac failure; Economics
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation | interventions — Digoxin; Ivabradine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Digoxin cross-over ivabradine: Digoxin 0,125 mg once a day 5 days per week during 3 months. Ivabradine, 7,5 mg b.id. during 3 months.
  Interventions: Drug: Digoxin and ivabradine

INTERVENTIONS:
Drug: Digoxin and ivabradine — No more details
  Other Names: Medical therapy in heart failure with atrial fibrillation.; Drugs used: digoxin and ivabradine.

SUMMARY:
This is an investigator-started study. The trial is coded as no. GC&PJ-Dig-Iva2009-2012.

The authors have no conflict of interest and there was no financial sponsoring The study was planned according to the Good Clinical Quality standards using an intention-to-treat analysis. The protocol was approved from the ethics committee. Selected patients gave their written informed consent. The family practitioners agreed and obtained the collected data and analysis. Analysis of collected data was performed by a single-blinded author (without knowledge of the used test drug and time of collection of data).

Study Hypothesis: Compare the effect of digoxin and ivabradine in chronic heart failure with permanent atrial fibrillation (ischemic etiology).

Multiple Time Frames: Primary Outcome is measured before and after each medical intervention.

Measurements at baseline and after 3 month of therapy (twice, with the 2 different drugs):

Measurements Severity of dyspnea. Digoxin serum concentration. ECG: Heart rate at rest and during 6-min walking test. Cardiac function (echocardiography): systolic function (ejection rate, left trial size,diastolic function.

Participants were followed (ambulatory observation) for at least 3 months

DETAILED DESCRIPTION:
Selected patients had chronic coronary artery disease which had been treated with percutaneous dilatation & stenting and/or aortocoronary bypass. The severity of myocardial ischemia had induced heart failure with diastolic dysfunction and preserved systolic function, and permanent AF.

1 Inclusion criteria:

Dyspnea class III NYHA.

Abnormal left ventricular relaxation with preserved (≥52%) ejection fraction (LVEF).

Patients either in sinus rhythm or with permanent atrial fibrillation.

2. Exclusion criteria:

Unstable angina pectoris.

Reduced systolic cardiac function (LVEF<52%).

Normal diastolic function.

Diabetes requiring insulin.

Moderate or severe renal or hepatic dysfunction.

Technically insufficient echocardiography.

ELIGIBILITY:
Inclusion Criteria:

No need to change concomitant pharmacological therapy in the following months, dyspnea class III NYHA, and abnormal left ventricular relaxation with preserved (≥52%) left ventricular ejection fraction (LVEF).

Exclusion Criteria:

Unstable myocardial ischemia, reduced systolic cardiac function (LVEF<52%), diabetes mellitus requiring insulin, moderate or severe renal or hepatic dysfunction, or technically insufficient echocardiography.

Ages: 60 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic heart disease and heart failure with preserved systolic function, dyspnea grade III NYHA. Either in sinus rhythm (and possible paroxismal atrial fibrillation) or with permanent atrial fibrillation.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2008-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Cardiac function (diastolic and systolic function) | After 12-14 weeks
  Cardiac function (echocardiography): systolic function (i.e. LVEF) and diastolic function (Doppler E/A ratio, tissue Doppler e/e1 ratio, Doppler deceleration time of the E wave.

SECONDARY OUTCOMES:
Heart rate and blood pressure. | After 12-14 weeks
  Changes in heart rate and blood pressure.
Dyspnea. | After 12-14.weeks
  Changes in dyspnea NYHA class).
NB-proBNP value | After 12-14 weeks
  Changes (serum values) after therapy.
Body weight | 12-14. weeks
  Changes after therapy
Left atrial size | After 12-14 weeks
  Change (size).
ECG | After 12-14 weeks
  Changes (heart rate,PR-interval, QRS morphology and duration), ST-T segment, other arrhythmias
Laboratory | After 12-14 weeks
  Any changes in hematology, electrolytes, renal and hepatic function.
Side-effects | After 12-14 weeks
  Any side-effects, spontaneously reported or after specific questionining.
6-min walk test | After 12-14 weeks.
  Changes in length of the walk test and heart rate during the test.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Cocco, MD, Principal Investigator — Cardiologist, senior lecturer
Locations (1):
- Cardiology office, Rheinfelden, Canton of Aargau, Switzerland

REFERENCES:
- [Result] Cocco G, Jerie P. Comparison of digoxin and ivabradine in heart failure with preserved systolic function. Submitted to the American Heart Journal.